CLINICAL TRIAL: NCT05093478
Title: The Prevalence of Local IgE Elevation and Its Effect on Intranasal Capsaicin Therapy in the Non-allergic Rhinitis Population
Brief Title: The Prevalence of Local Immunoglobulin E (IgE) Elevation and Its Effect on Intranasal Capsaicin Therapy in the Non-allergic Rhinitis Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: American Academy of Otolaryngic Allergy (Other)
Responsible Party: Principal Investigator, Kunal R. Shetty, Otolaryngology Resident, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-19-0333
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Non-allergic Rhinitis
Keywords: rhinorrhea; congestion; sneezing; itching
MeSH Terms: conditions — Common Cold; Rhinorrhea; Sneezing; Pruritus | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Intranasal capsaicin; Drug: topical lidocaine

INTERVENTIONS:
Drug: Intranasal capsaicin — Intranasal capsaicin, 5 applications each delivering 2 micrograms in each nostril, separated by 1 hour.
Drug: topical lidocaine — The nose will be pre-treated with topical lidocaine 15 minutes before each application

SUMMARY:
The purpose of this study to determine the therapeutic response of non-allergic rhinitis patients that have been subtyped as non-allergic rhinitis with local IgE elevation or non-allergic rhinopathy to intranasal capsaicin based on visual analog scale and optical rhinometry, to determine the prevalence of non-allergic rhinitis with local IgE elevation in this study's cohort of patients with non-allergic rhinitis identified by rhinitis history and negative skin testing for allergic rhinitis, and to determine the change, if any, in intranasal IgE levels after capsaicin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic rhinitis

Exclusion Criteria:

* Active smoker
* Anatomic source of nasal symptoms
* Chronic rhinosinusitis or other nasal infection
* History of sinonasal malignancy
* Pregnancy or lactation
* Use of medication affecting nasal function (topical steroids, topical anticholinergics, oral antihistamines) in the previous 4 weeks
* Use or abuse of nasal decongestants.
* Positive skin prick test for allergic rhinitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kunal R Shetty, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 28
Completed | 24
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not collected from one participant in the treatment arm.
  years
    number analyzed (Participants) | 27
    (all) | 62.59 (16.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Runny Nose as Measured by the Visual Analog Scale (VAS) at Baseline
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 28
score on a scale | 6.07 (2.41)

2. Primary Outcome: Runny Nose as Measured by the Visual Analog Scale (VAS) at 4 Weeks Post Treatment
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: 4 weeks post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 28
score on a scale | 2.89 (2.04)

3. Primary Outcome: Runny Nose as Measured by the Visual Analog Scale (VAS) at 12 Weeks Post Treatment
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: 12 weeks post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 24
score on a scale | 3.75 (3.15)

4. Primary Outcome: Nasal Symptoms of Congestion as Measured by the Visual Analog Scale (VAS) at Baseline
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 28
score on a scale | 5.57 (2.80)

5. Primary Outcome: Nasal Symptoms of Congestion as Measured by the Visual Analog Scale (VAS) at 4 Weeks Post Treatment
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: 4 weeks post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 28
score on a scale | 2.46 (2.13)

6. Primary Outcome: Nasal Symptoms of Congestion as Measured by the Visual Analog Scale (VAS) at 12 Weeks Post Treatment
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: 12 weeks post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 24
score on a scale | 2.75 (2.13)

7. Primary Outcome: Nasal Itching as Measured by the Visual Analog Scale (VAS at Baseline
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 28
score on a scale | 2.25 (2.60)

8. Primary Outcome: Nasal Itching as Measured by the Visual Analog Scale (VAS) at 4 Weeks Post Treatment
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: 4 weeks post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 28
score on a scale | 1.50 (1.95)

9. Primary Outcome: Nasal Itching as Measured by the Visual Analog Scale (VAS) at 12 Weeks Post Treatment
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: 12 weeks post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 24
score on a scale | 1.20 (1.84)

10. Primary Outcome: Nasal Sneezing as Measured by the Visual Analog Scale (VAS) at Baseline
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 28
score on a scale | 3.03 (2.47)

11. Primary Outcome: Nasal Sneezing as Measured by the Visual Analog Scale (VAS) at 4 Weeks Post Treatment
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: 4 weeks post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 28
score on a scale | 1.71 (2.07)

12. Primary Outcome: Nasal Sneezing as Measured by the Visual Analog Scale (VAS) at 12 Weeks Post Treatment
Description: The Visual analog scale is scored from 0-10, with 0 being not a problem and 10 being unbearable.
Time Frame: 12 weeks post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 24
score on a scale | 2.29 (2.91)

13. Primary Outcome: Change in Maximum Optical Density Determined Via Optical Rhinometry
Description: Optical rhinometry provides continuous measurement of blood flow in nasal vessels (via optical density measurements), which serves as an indirect assessment of nasal congestion. A greater decrease in optical density (OD) from baseline indicates less nasal blood flow and decreased congestion relative to baseline.
Time Frame: baseline, immediately post first treatment on Day 1
Population: Data were not collected for 6 participants in the treatment arm.
Measure: Mean (Standard Deviation); unit: log ratio of light in to light out (OD)
Arm/Group | Treatment
Number analyzed (Participants) | 22
log ratio of light in to light out (OD) | 0.36 (0.18)

14. Primary Outcome: Total Nasal Symptom Score as Measured by the Visual Analog Scale (VAS) at Baseline
Description: Total Nasal Symptom score is measured as the sum of four symptom scores for runny nose, nasal symptoms of congestion, nasal itching and sneezing. Each symptom is scored from 0-10, with 0 being not a problem and 10 being unbearable. The Total nasal symptom score ranges from 0 - 40, the lower the score the better the outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 28
score on a scale | 16.92 (7.03)

15. Primary Outcome: Total Nasal Symptom Score as Measured by the Visual Analog Scale (VAS) at 4 Weeks Post Treatment
Description: as for outcome 14
Time Frame: 4 weeks post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 28
score on a scale | 8.57 (6.69)

16. Primary Outcome: Total Nasal Symptom Score as Measured by the Visual Analog Scale (VAS) at 12 Weeks Post Treatment
Description: as for outcome 14
Time Frame: 12 weeks post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 24
score on a scale | 10 (7.78)

17. Secondary Outcome: Change in Local Immunoglobulin E (IgE) Level
Description: The IgE levels will be obtained from the brush biopsy of the inferior turbinates. Change from baseline in local Immunoglobulin E (IgE) level after 12 weeks post treatment. Data reported is the 12 weeks post treatment value minus the baseline value.
Time Frame: baseline, 12 weeks post treatment
Population: Data were not collected for 5 participants in the Treatment arm.
Measure: Mean (Standard Deviation); unit: kU/L
Arm/Group | Treatment
Number analyzed (Participants) | 19
kU/L | 0.17 (1.57)

18. Primary Outcome: Maximum Optical Density Determined Via Optical Rhinometry
Time Frame: 12 weeks post treatment
Population: Data were not collected for this outcome measure.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT05093478/Prot_SAP_000.pdf